CLINICAL TRIAL: NCT05930548
Title: Clinical Evaluation of Low-shrinkage Giomer Resin Composite Versus Resin-Modified Glass Ionomer in Treatment of Cervical Caries Lesions: A Randomized Clinical Trial
Brief Title: Evaluation of Low-shrinkage Giomer Versus Resin-Modified Glass Ionomer in Cervical Caries Lesions: A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Menna Omar El Ghamrawy, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSG_RMGI
Record Dates: First submitted 2023-06-23; First posted 2023-07-05 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Caries, Cervical
Keywords: Cervical carious lesions; Low shrinkage giomer resin composite; Resin modified glass ionomer; FDI criteria
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resin modified glass ionomer (Active Comparator): RMGI is recommended to restore carious cervical lesions; especially with its ability to inhibit secondary caries due to its fluoride releasing ability. The main advantage of RMGI is its capability to chemically bond to tooth structure, even in the presence of moist dentin. RMGI reaction can be achieved by both acid-base reaction (induced by glass ionomer component) and polymerization reaction (induced by resin component). Thus, RMGI has better mechanical properties, wear resistance, and improved esthetics compared with conventional glass ionomer (AlQranei MS et al, 2021). In addition, the coefficient of thermal expansion of glass ionomer which is similar to that of tooth structure, allows for proper marginal adaptation without marginal leakage (Bollu IP et al, 2016).
  Interventions: Other: Low Shrinkage Giomer
- Low shrinkage giomer (Experimental): Low shrinkage giomer resin composite shows both sustained fluoride release and recharge, and low volumetric shrinkage of less than 1% with low resultant polymerization shrinkage stress. Such remarkable feature is due to the novel SRS (Steric Repulsion Structured) molecule which is designed to decrease polymerization shrinkage through molecular steric repulsion resulting in a stable restoration microstructure (AlQranei MS et al, 2021). Thus, low shrinkage giomers are best indicated in class V cavities where the dentin bonding agent does not have high strength (Algailani U, et al 2022).
  Interventions: Other: Low Shrinkage Giomer

INTERVENTIONS:
Other: Low Shrinkage Giomer — Low shrinkage giomer resin composite shows both sustained fluoride release and recharge, and low volumetric shrinkage of less than 1% with low resultant polymerization shrinkage stress. Such remarkable feature is due to the novel SRS (Steric Repulsion Structured) molecule which is designed to decrease polymerization shrinkage through molecular steric repulsion resulting in a stable restoration microstructure (AlQranei MS et al, 2021). Thus, low shrinkage giomers are best indicated in class V cavities where the dentin bonding agent does not have high strength (Algailani U, et al 2022).

SUMMARY:
Management of cervical lesions presents serious problems with any restorative material. The two most common reasons for restoration failure are secondary caries at the tooth-restoration interface and loss of retention. Class V lesions often exhibit a low retentive cavity configuration (C-factor); which is responsible for marginal gaps around the restorations. Cervical margins -lying in either dentin or cementum- show unfavorable bonding performance, besides being usually subgingival where moisture control is difficult. The subgingival margin is not clinically desirable due to difficulty in cleaning and increased biofilm accumulation. Therefore, the selection of the restorative material can be challenging.

Resin composites are known for their high mechanical properties, excellent esthetic properties, and ease of clinical application. However, when compared with glass ionomers, resin composite has no cariostatic effect on tooth structure. In addition, microleakage caused by polymerization shrinkage of resin composite leads to plaque accumulation and secondary caries. On the other hand, resin-modified glass ionomer has many advantages, yet still it has lower weakness and esthetic properties compared to resin composite.

Based on current literature, there is limited evidence comparing clinical performance of low-shrinkage giomer resin composite to resin-modified glass ionomer in the treatment of cervical caries lesions.

This study is conducted to evaluate the clinical performance of low-shrinkage giomer resin composite versus resin-modified glass ionomer in treatment of cervical caries lesions, using both Modified USPHS and Revised FDI criteria. This study will be designed to test the null hypothesis that the low-shrinkage giomer resin composite will have the same clinical performance as resin-modified glass ionomer in cervical restorations, using both Modified USPHS and Revised FDI criteria.

DETAILED DESCRIPTION:
The development of cervical lesions in permanent dentition may be related to carious or non- carious origin. Class V caries lesions may occur due to different factors such as poor oral hygiene, dietary habits, or xerostomia.

Management of cervical lesions presents serious problems with any restorative material. The two most common reasons for restoration failure are secondary caries at the tooth-restoration interface and loss of retention. Class V lesions often exhibit a low retentive cavity configuration (C-factor); which is responsible for marginal gaps around the restorations. Cervical margins -lying in either dentin or cementum- show unfavorable bonding performance, besides being usually subgingival where moisture control is difficult. The subgingival margin is not clinically desirable due to difficulty in cleaning and increased biofilm accumulation. Therefore, the selection of the restorative material can be challenging.

In this context, fluoride containing adhesive materials are considered ideal in restoring class V carious lesions. Resin modified glass ionomers (RMGI) are highly recommended in the restoration of cervical lesions. The most important advantages of glass ionomer are its chemical adhesion to the tooth structure, and its fluoride release. However, RMGI has lower weakness and esthetic properties compared to resin composite.

In our study, the comparator material will be light cured resin reinforced glass ionomer restorative. RMGI is recommended to restore carious cervical lesions; especially with its ability to inhibit secondary caries due to its fluoride releasing ability. The main advantage of RMGI is its capability to chemically bond to tooth structure, even in the presence of moist dentin. RMGI reaction can be achieved by both acid-base reaction (induced by glass ionomer component) and polymerization reaction (induced by resin component). Thus, RMGI has better mechanical properties, wear resistance, and improved esthetics compared with conventional glass ionomer. In addition, the coefficient of thermal expansion of glass ionomer which is similar to that of tooth structure, allows for proper marginal adaptation without marginal leakage.

Resin composites have been widely used in dental practice; because of their high mechanical properties, excellent esthetic properties, and ease of clinical application.

However, when compared with glass ionomers, resin composite has no cariostatic effect on tooth structure. In addition, polymerization shrinkage of resin composite is of major concern; where mechanical stresses are developed due to contraction leading to break the marginal seal between resin composite and tooth structure. Polymerization shrinkage can cause clinical issues as restoration or tooth fracture, bond degradation and solubility, and microleakage. The microleakage caused by polymerization shrinkage of resin composite leads to plaque accumulation and secondary caries. Thus, choosing a fluoride-releasing and low-shrinkage resin composite may play a critical role in success of cervical restorations.

The continued development of resin composites has led to the introduction of Giomer technology. By combining the characteristics of resin composite and glass ionomer, hybrid products called giomers have been obtained. Giomer resin composite offers protection against caries, along with improved functional and esthetic properties; through incorporating particles of pre-reacted glass fillers (PRG) into the matrix of resin composite. The PRG-ionomer phase has the capability to release six key ions which are fluoride, aluminum, borate, silicate, strontium, and sodium ions. These ions exhibit acid neutralizing ability and help prevent demineralization of enamel and dentin, leading to decrease the possible incidence of secondary caries. This PRG technology provides giomer with both fluoride release and recharge, similar to glass ionomer while still maintaining the original physical properties of resin composite.

Beautifil™ II LS (Low shrinkage) giomer resin composite (Shofu Inc, Kyoto, Japan) shows both sustained fluoride release and recharge, and low volumetric shrinkage of less than 1% with low resultant polymerization shrinkage stress. Such remarkable feature is due to the novel SRS (Steric Repulsion Structured) molecule which is designed to decrease polymerization shrinkage through molecular steric repulsion resulting in a stable restoration microstructure. Thus, low shrinkage giomers are best indicated in class V cavities where the dentin bonding agent does not have high strength.

A recent clinical trial compared the clinical performance of giomers versus resin modified glass ionomer in proximal lesions. Marginal adaptation was higher in giomers than resin-modified glass ionomers after 12 months. Also, a systematic review investigated in vivo longevity of giomers compared to other adhesive restorative materials (hybrid resin composite, composmer, and RMGIC), and concluded that RMGIC was the most successful material in terms of biological properties while giomers had the longest survival rate. An in-vitro study evaluated the surface roughness and fluoride release of Beautifil II and Fuji II LC (resin-modified glass ionomer). Resin-modified glass ionomer showed the highest fluoride release, while the giomer showed an intact, smooth surface with no irregularities as those found in glass ionomer. Thus, the smooth surface of giomers inhibit biofilm formation, decreasing the risk of dental caries and periodontal diseases. Regarding the mechanical properties of giomers, it has exhibited a higher flexural strength value when compared to glass ionomer cements. The hardness values were twice as high for the giomer when compared to self-curing and light-curing glass ionomer cements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carious cervical lesions in maxillary anterior teeth. Patients with at least 20 teeth under occlusion.
* Age: 25-50 years.
* Males or females
* Asymptomatic vital teeth. No pulp pathology or periapical pathosis
* Healthy periodontium and favorable occlusion.
* Good general health
* Co-operative patients approving to participate in the trial.

Exclusion Criteria:

* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.
* Parafunctional habits or TMJ disorders
* Active periodontitis
* Teeth supporting removable prostheses, or orthodontic appliances.
* Candidates with parafunction or bruxism.
* Candidates with systemic diseases or disabilities that may affect participation.
* Xerostomia.
* Heavy smoking.
* Pregnancy.
* Lack of compliance.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Clinical performance | 12 months: change from baseline to six, and 12 months.
  fracture and retention, marginal adaptation, form and contour, caries at the restoration margins, dental hard tissue defects, and postoperative hypersensitivity, surface luster and surface texture, marginal staining, and color match All these outcomes are measured using revised FDI criteria for clinical evaluation of restoration; where they will be given a score either excellent (1), good (2), satisfactory (3), unsatisfactory (4), or poor (5) - (acceptable = score 1 to 3, inacceptable but repair possible = score 4, and inacceptable but repair not possible/reasonable = score 5).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Giza, Egypt

REFERENCES:
- [Derived] El Ghamrawy M, Kamal D, Hamza H. Clinical performance and cost-effectiveness of low-shrinkage giomer resin composite versus resin-modified glass ionomer in cervical carious lesions: a 12-month randomized controlled trial. BMC Oral Health. 2025 Aug 6;25(1):1295. doi: 10.1186/s12903-025-06594-y. PMID 40770630

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT05930548/Prot_SAP_ICF_000.pdf